CLINICAL TRIAL: NCT03749031
Title: The Effect of Orange or Apple Pomace on Digestive Health in Adults: a Randomized, Double Blind, Controlled Trial
Brief Title: Effects of Beverages Containing Orange or Apple Pomace on Digestive Health in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1805
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Digestive Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Orange juice only (Placebo Comparator): 16 oz. orange juice per day for 4 weeks
  Interventions: Other: Orange Juice
- orange juice + orange Pomace (Experimental): 16 oz. orange juice + orange Pomace per day for 4 weeks
  Interventions: Other: Orange juice + Orange Pomace
- Apple juice only (Placebo Comparator): 16 oz. apple juice per day for 4 weeks
  Interventions: Other: Apple Juice
- Apple Juice + Apple Pomace (Experimental): 16 oz. apple juice + apple Pomace per day for 4 weeks
  Interventions: Other: Apple Juice and Apple Pomace

INTERVENTIONS:
Other: Orange juice + Orange Pomace — 16 oz. orange juice + orange Pomace per day for 4 weeks
  Arms: orange juice + orange Pomace
Other: Orange Juice — 16 oz. orange juice per day for 4 weeks
  Arms: Orange juice only
Other: Apple Juice and Apple Pomace — 16 oz. apple juice and apple Pomace per day for 4 weeks
  Arms: Apple Juice + Apple Pomace
Other: Apple Juice — 16 oz. apple juice per day for 4 weeks
  Arms: Apple juice only

SUMMARY:
This is a randomized crossover intervention designed to evaluate effects of daily intake of beverages containing orange or apple Pomace on gastrointestinal function as measured by stool frequency. Additional outcomes will include aspects of digestive health and self-reported GI symptoms and dietary intake as well as analysis of gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females 18-60 years old
* Willing and able to consume 16 oz. of orange or apple beverage per day for 4 week periods
* Willing to maintain usual diet, smoking status, physical activity pattern, supplements and meds

Exclusion Criteria:

* Food allergies or sensitivities to ingredients in study beverages
* Presence or history of GI condition, endocrine (including diabetes), cardiovascular disease or other disease or condition that could interfere in the interpretation of the study results in the opinion of the Investigator.
* Extreme dietary habits including vegetarian, vegan or Atkins diet
* Females or are pregnant, planning to become pregnant or breast feeding during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
stool frequency | Changes over 7 weeks (daily during 4 week treatment followed by daily during 3 week washout) compared to baseline (daily during 2 week run-in)
  Bowel habits daily diary as weekly averages. Fewer days with no stool, and higher number of stools per week would be better.

SECONDARY OUTCOMES:
Self-reported GI symptoms | Changes over 7 weeks (daily during 4 week treatment followed by daily during 3 week washout) compared to baseline (daily during 2 week run-in)
  GI Tolerability questionnaire, 4 selections. The minimum value is Less than usual. The maximum value is Much more than usual. Pomace treament arms expected to have more GI symptoms than juice arms. Less symptoms are better than more.
Stool consistency | Changes over 7 weeks (daily during 4 week treatment followed by daily during 3 week washout) compared to baseline (daily during 2 week run-in)
  Bristol score, 7 types of stool drawings presented in a chart from lumpy Type 1, to watery Type 7. Improved consistency would be better.
Ease of stool passage | Changes over 7 weeks (daily during 4 week treatment followed by daily during 3 week washout) compared to baseline (daily during 2 week run-in)
  Rating scale 1 (Very easy) to 5 (Very difficult). Easier passage would be better.
microbiota changes | Changes from baseline sample to end of treatment sample (Week 4) and end of 3 week washout sample (Week 7)
  Stool samples for possible explanations of mechanisms of pomace. Higher bacteria associated with fiber fermentation would be better. Species examined include F. Prau, lachnospiraceae, ruminoucoccaceae, bifidobacteria, and changes in alpha and beta diversity as measured by 16S RNA sequencing. Data pending, unknown units at this time.
Dietary analysis | Changes from 2 week run in (baseline) to the last week of treatment (Week 4) and the last week of 3 week washout (Week 7)
  3-day diet record. Expecting higher daily fiber intake for pomace arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, MD, Principal Investigator — BioFortis
Locations (1):
- BioFortis, Addison, Illinois, United States